CLINICAL TRIAL: NCT06131658
Title: Effects of Functional Motor Control Exercise on Pain, Flexibility, Lower Extremity Function Among Runners With Iliotibial Band Syndrome
Brief Title: Effects of Functional Motor Control on Pain, Flexibility, Lower Extremity Function With ITBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0429
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Iliotibial Band Syndrome; Pain; Flexibility
Keywords: motor control function excercise; lower extermity function; Iliotibial Band Syndrome
MeSH Terms: conditions — Iliotibial Band Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: assessor who will take reading is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional motor control excercise (Experimental): Functional motor control exercise Includes side plank with clamshell, Side plank with hip abduction, Side-lying hip abduction, Lateral monster walk, Hip hikes, Single leg squat, TKE with T-band-hip abduction All exercises done with 2 sets of 10 reps with 3 sessions per week for 6 weeks
  Interventions: Other: Functional motor control excercise
- conventional exercise (Experimental): The conventional exercise included 4 stages of self-myofascial techniques, strengthening, and integration techniques. In the first phase, individuals did fascial release exercises using foam rolls, focusing on tensor fascia latae, iliotibial band, and hip adductor muscles, and tennis balls for the quadratus lumborum. The exercises were performed at high-intensity maximum pain tolerance for 30 seconds or low-intensity minimum pain tolerance for 90 seconds.
  Interventions: Other: convectional excercise

INTERVENTIONS:
Other: Functional motor control excercise — This include functional motor control thrice a week for six weeks
  Arms: Functional motor control excercise
Other: convectional excercise — This include convectional exercise thrice a week for six weeks
  Arms: conventional exercise

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by non-probability convenient random sampling technique. Subjects in group A will receive functional motor control exercises. Group B will receive conventional exercises.

DETAILED DESCRIPTION:
The objective of this study is to determine the effects of functional motor control exercises on pain, flexibility and lower limb functional. It will be randomized controlled trial (RCT) research design at Pakistan sports board through non probability convenience sampling technique on 72 runners' athletes which will be allocated using random sampling through computerized generated number into Group A and Group B, 36 athletes will be in each group. Group A (interventional) will be given conventional training with functional motor exercise and Group B (control) will be given conventional training. There will be 3 sessions in a week for 6 weeks. The baseline scoring will be on 1st day, follow up will be taken at 6th week. Assessment will be made by Numeric pain rating scale, Lower extremity functional scale (LEFS), Single leg mini squat, Y balance. Data will be analyzed during SPSS software version 26. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two group

ELIGIBILITY:
Inclusion Criteria:

* male and female athlete within 19-40 years,
* running a minimum average of 15 running kilometers,
* Runners with one sided iliotibial band syndrome for at least 3 months were included,
* Pain along IT band at either Gerdy's tubercle or the lateral femoral epicondyle during running,
* positive stiffness with Ober's test, and
* reporting pain during Noble's compression test.

Exclusion Criteria:

* Individuals with a history of previous knee trauma of past 6 months,
* Individuals with a history of previous knee surgery of past 6 months,
* Other knee abnormalities including patellofemoral joint pain,
* popliteus tendinitis,
* lateral meniscal injury,
* Degenerative joint disease, and
* lateral collateral ligament sprain to the affected side.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | pre and 6 weeks post interventional
  pain will be assess by Numeric pain rating scale with minimum score 0 to maximum score 10
flexibility | pre and 6 weeks post interventional
  flexibility will be assess by Y balance
lower extremity function | pre and 6 weeks post interventional
  lower extremity function will be assess by lower limb extremity scale with score 0 to 80

CONTACTS AND LOCATIONS:
Overall Officials: maham Athar, DPT, Principal Investigator — Investigator
Locations (1):
- Jawad Club, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKean KA, Manson NA, Stanish WD. Musculoskeletal injury in the masters runners. Clin J Sport Med. 2006 Mar;16(2):149-54. doi: 10.1097/00042752-200603000-00011. PMID 16603885
- [Background] Taunton JE, Ryan MB, Clement DB, McKenzie DC, Lloyd-Smith DR, Zumbo BD. A retrospective case-control analysis of 2002 running injuries. Br J Sports Med. 2002 Apr;36(2):95-101. doi: 10.1136/bjsm.36.2.95. PMID 11916889
- [Background] Fredericson M, Cookingham CL, Chaudhari AM, Dowdell BC, Oestreicher N, Sahrmann SA. Hip abductor weakness in distance runners with iliotibial band syndrome. Clin J Sport Med. 2000 Jul;10(3):169-75. doi: 10.1097/00042752-200007000-00004. PMID 10959926
- [Background] Baker RL, Fredericson M. Iliotibial Band Syndrome in Runners: Biomechanical Implications and Exercise Interventions. Phys Med Rehabil Clin N Am. 2016 Feb;27(1):53-77. doi: 10.1016/j.pmr.2015.08.001. PMID 26616177
- [Background] Noehren B, Davis I, Hamill J. ASB clinical biomechanics award winner 2006 prospective study of the biomechanical factors associated with iliotibial band syndrome. Clin Biomech (Bristol). 2007 Nov;22(9):951-6. doi: 10.1016/j.clinbiomech.2007.07.001. Epub 2007 Aug 28. PMID 17728030